CLINICAL TRIAL: NCT05694741
Title: A Phase 1 Randomized, Single-blind, Placebo-controlled, First-in-Human and Sequential Group Study to Assess Safety, Tolerability, and Pharmacokinetics of AZD0186 Following Single Ascending Doses Via Oral Administration
Brief Title: A Study to Assess Safety, Tolerability, and Pharmacokinetics of AZD0186
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision was based on the overall data profile obtained from this study which did not demonstrate sufficient differentiation to surpass the current standard of care.
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: D8740C00001
Record Dates: First submitted 2022-12-20; First posted 2023-01-23 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Hyperglycemia; Glucagon-like peptide-1 receptor agonists
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia

STUDY DESIGN:
Intervention Model Description: Placebo-control
Who Masked: Care Provider, Investigator
Masking Description: Sponsor-open
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (healthy volunteers) (Experimental): The planned number of cohorts is up to 6 cohorts; additional cohorts may be included if it is considered necessary to repeat a dose level or if additional dose steps are required for safety purposes. Six subjects will receive AZD0186, and two subjects will receive placebo.
  Interventions: Drug: AZD0186; Drug: Placebo
- Cohort 2 (healthy Japanese volunteers) (Experimental): The planned number of Japanese cohorts is 1, but more than 1 cohort may be included if the SRC considers it necessary to repeat a dose level or if additional dose steps are required. No sentinel dosing will be performed for the Japanese cohort.
  Interventions: Drug: AZD0186; Drug: Placebo
- Cohort 3 (healthy Chinese volunteers) (Experimental): The planned number of Chinese cohorts is 1, but more than 1 cohort may be included if it is considered necessary to repeat a dose level or if additional dose steps are required. No sentinel dosing will be performed for the Chinese cohort.
  Interventions: Drug: AZD0186; Drug: Placebo
- Cohort 4 (healthy volunteers - food effect) (Experimental): One of the Part 1 cohorts (planned for Cohort 6, can be updated pending emerging data) will continue into the food-effect part after a washout period. This part will be initiated after SRC review of all available data from preceding cohorts in this study.
  Interventions: Drug: AZD0186; Drug: Placebo

INTERVENTIONS:
Drug: AZD0186 — Subjects will receive AZD0186 orally.
Drug: Placebo — Subjects will receive placebo orally.

SUMMARY:
This study will assess the safety, tolerability, and pharmacokinetics of AZD0186 following single ascending doses (SAD) via oral administration in healthy adult participants.

DETAILED DESCRIPTION:
This is a Phase 1, First-in-Human (FIH), randomized, single-blind, sponsor-open, placebo-controlled, SAD sequential group design study.

This study consists of four parts: Part 1, Part 2, Part 3, and Part 4.

The study will comprise of the following:

Part 1, Part 2, Part 3, and Part 4:

* A Screening Period of maximum 28 days.
* A Treatment Period during which subjects will be resident at the Clinical Unit from 2 days before IMP (Investigational Medicinal Product) administration (Day -2) until at least 48 hours after IMP administration; discharged on Day 3.

Part 4:

• A second Treatment Period during which subjects will be resident at the Clinical Unit from the day of the Follow-up Visit (Day 7 ±1 days after the last IMP dose) until at least 48 hours after the second IMP administration; discharged on Day 10.

Part 1, Part 2, Part 3, and Part 4:

• A Follow-up Visit after 7 (Part 1, Part 2, and Part 3) or 14 (Part 4) ±1 day after the last IMP dose.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy male and female subjects aged 18 to 55 years with suitable veins for cannulation or repeated venipuncture.
* Females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit, must not be lactating and must be of non-childbearing potential, confirmed at the Screening Visit.
* Have a BMI between:

  1. Part 1: 18 to 32 kg/m2 inclusive,
  2. Part 2 and Part 3: 18 to 32 kg/m2 inclusive,
  3. and weigh at least 50 kg (males and females).
* Provision of signed, written, and dated informed consent for optional genetic/biomarker research.
* For the healthy Japanese cohort (Part 2): healthy subjects are to be Japanese (eg, natives of Japan or Japanese Americans), defined as having both parents and 4 grandparents who are Japanese.
* For the healthy Chinese cohort (Part 3): healthy male and female (of non-childbearing potential) healthy Chinese subjects for whom both parents and all grandparents are Chinese and not lived outside of China for more than 10 years.

Exclusion Criteria:

* History of any clinically important disease or disorder which may either put the healthy subject at risk because of participation in the study,or influence the results or the healthy subject's ability to participate in the study.
* History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
* Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP.
* Presence of any retinal (including intraretinal) abnormality detected by ophthalmological examination including indirect ophthalmoscopy, fundoscopy or OCT.
* Presence of any factors that predispose to retinal detachment including lattice degeneration, retinal hole, or high myopia (-10 diopters or higher) found on ophthalmological examination.
* History of retinal detachment in either eye.
* History of treated or untreated retinal holes.
* Any clinically important abnormalities across the ophthalmological examinations.
* Any laboratory values with the following deviations:

  1. Alanine aminotransferase > ULN
  2. Aspartate aminotransferase > ULN
  3. eGFR < 90 mL/minute/1.73 m2 (calculated using the Chronic Kidney Disease Epidemiology Collaboration formula)
  4. White blood cell count < LLN
  5. Hemoglobin < LLN
* Any clinically important abnormalities in clinical chemistry, hematology or urinalysis results.
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody and HIV.
* Abnormal vital signs, after 10 minutes supine rest, defined as any of the following:

  1. Systolic BP < 90 mmHg or > 140 mmHg.
  2. Diastolic BP < 50 mmHg or > 90 mmHg.
  3. Heart rate < 45 or > 85 bpm.
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting ECG and any clinically important abnormalities in the 12-lead ECG that may interfere with the interpretation of QTc interval changes, including abnormal ST and T-wave morphology, particularly in the protocol defined primary lead or left ventricular hypertrophy.
* Known or suspected history of drug abuse.
* Current smokers or those who have smoked or used nicotine products within the previous 3 months.
* History of alcohol abuse or excessive intake of alcohol.
* Positive screen for drugs of abuse or cotinine at screening or admission to the Clinical Unit or positive screen for alcohol on admission to the Clinical Unit prior to the first administration of the IMP.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to GLP-1 RA.
* Any condition that would have interfered with the evaluation of the IMP or interpretation of subject safety or study results.
* Lifetime history of schizophrenia or other psychosis or bipolar disorder or suicide attempts, major depressive disorder, or self-reported suicidal ideation.
* Healthy subjects with a history of MTC, multiple endocrine neoplasia syndrome type 2, or healthy subjects with a screening/baseline serum calcitonin ≥ 50 pg/mL.
* History of gastrointestinal abnormality that could affect gastrointestinal motility.
* Excessive intake of caffeine containing drinks or food.
* Plasma donation within one month of the Screening Visit or any blood donation/blood loss > 500 mL during the 3 months prior to the Screening Visit.
* Has received another new chemical entity within 30 days or 5 half-lives of the first administration of IMP in this study.
* Previous bone marrow transplant.
* Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs), and Serious Adverse Events (SAEs) | Up to the Follow-up Visit (approximately 6 weeks)
  The safety and tolerability of AZD0186 following oral single ascending doses in healthy subjects (Part 1 and Part 4), in healthy Japanese subjects (Part 2), and in healthy Chinese subjects (Part 3) will be assessed.

SECONDARY OUTCOMES:
Area under plasma concentration-time curve from zero to infinity (AUCinf) | Day 1 to Day 3
  The AUCinf of AZD0186 following oral single ascending doses will be characterized.
Area under the plasma concentration-time curve from 0 to the last quantifiable concentration (AUClast) | Day 1 to Day 3
  The AUClast of AZD0186 following oral single ascending doses will be characterized.
Maximum observed concentration (Cmax) | Day 1 to Day 3
  The Cmax of AZD0186 following oral single ascending doses will be characterized.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Yoon, MD, Principal Investigator — PAREXEL Early Phase Clinical Unit-Los Angeles
Locations (1):
- Research Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual participant-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: D8740C00001_Redacted_CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8740C00001&attachmentIdentifier=a506b377-16f9-445b-bb42-6620c0728261&fileName=D8740C00001_Redacted_CSR_Synopsis.pdf&versionIdentifier=
- See also: D8740C00001_link to the results already presented on AZCT — https://www.astrazenecaclinicaltrials.com/study/D8740C00001/